CLINICAL TRIAL: NCT01077713
Title: Randomised Phase II Trial of Bevacizumab (AVASTIN®) in Combination With Gemcitabine or Attenuated Doses of Cisplatin and Gemcitabine as First-line Treatment of Elderly Patients With Advanced Non-squamous Non-small Cell Lung Cancer - EAGLES
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Gemcitabine With or Without Cisplatin in First-Line Treatment of Elderly Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21868; 2008-008739-27
Record Dates: First submitted 2010-02-09; First posted 2010-03-01 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Bevacizumab; Cisplatin; Gemcitabine

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: gemcitabine
- 2 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: cisplatin; Drug: gemcitabine

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 7.5mg/kg iv on day 1 of each 3 week cycle
Drug: cisplatin — 60mg/m2 on day 1 of each 3 week cycle
  Arms: 2
Drug: gemcitabine — 1200mg/m2 on days 1-8 of each 3 week cycle
  Arms: 1
Drug: gemcitabine — 1000mg/m2 on days 1-8 of each 3 week cycle
  Arms: 2

SUMMARY:
This 2 arm study will evaluate the efficacy and safety of Avastin + gemcitabine, and Avastin + gemcitabine + attenuated doses of cisplatin, as first line treatment in elderly patients with non-squamous non-small cell lung cancer. Patients will be randomised to receive either Avastin 7.5mg/kg iv on day 1 + gemcitabine 1200mg/m2 on days 1-8 of each 3 week cycle, or Avastin 7.5mg/kg iv on day 1 + cisplatin 60mg/m2 on day 1 + gemcitabine 1000mg/m2 on days 1-8 of each 3 week cycle. After 6 cycles of combination therapy, all patients will continue to receive Avastin monotherapy. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=70 years of age;
* inoperable, locally advanced, metastatic non-squamous non-small cell lung cancer;
* >=1 measurable lesion;
* ECOG performance status 0-1.

Exclusion Criteria:

* neoadjuvant/adjuvant chemotherapy within 6 months prior to enrollment;
* radical radiotherapy with curative intent within 28 days prior to enrollment;
* history of >=grade 2 hemoptysis in 3 months prior to enrollment;
* evidence of CNS metastases;
* current or recent (within 10 days of first dose of Avastin)use of aspirin (>325 mg/day)or full dose anticoagulants or thrombolytic agents for therapeutic purposes.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- Italy (24):
  - Rionero in Vulture, Basilicate
  - Catanzaro, Calabria
  - Avellino, Campania
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Aviano, Friuli Venezia Giulia
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Viterbo, Lazio
  - Genoa, Liguria
  - Bergamo, Lombardy
  - Milan, Lombardy
  - Monza, Lombardy
  - Rho, Lombardy
  - Sondalo, Lombardy
  - Sondrio, Lombardy
  - Novara, Piedmont
  - Catania, Sicily
  - Ancona, The Marches
  - Pesaro, The Marches
  - Lido di Camaiore, Tuscany
  - Perugia, Umbria
  - Mirano, Veneto
  - Padua, Veneto

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Gemcitabine: Participants received bevacizumab 7.5 milligrams per kilogram (mg/kg) intravenous (IV) infusion on Day 1 and gemcitabine 1200 milligrams per square meter (mg/m^2) IV infusion on Days 1 and 8 of each 21-day cycle for a maximum of 6 cycles. After Cycle 6, participants continued treatment with bevacizumab 7.5 mg/kg IV infusion on Day 1 of every 21-day cycle until progressive disease, death, or intolerable toxicity.
- Bevacizumab + Gemcitabine + Cisplatin: Participants received bevacizumab 7.5 mg/kg IV infusion and cisplatin 60 mg/m^2 IV infusion on Day 1 and gemcitabine 1000 mg/m^2 IV infusion on Days 1 and 8 of each 21-day cycle for a maximum of 6 cycles. After Cycle 6, participants continued treatment with bevacizumab 7.5 mg/kg IV infusion on Day 1 of every 21 day cycle until progressive disease, death, or intolerable toxicity.
Period: Overall Study
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Started | 44 | 42
Completed | 8 | 6
Not Completed | 36 | 36
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Progressive Disease (PD) | 0 | 1
Not completed — Death | 28 | 29
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Other | 4 | 2

BASELINE CHARACTERISTICS:
Population: All participants randomized set (RND) included all participants who provided informed consent and who were randomized to study medication.
Groups:
- Bevacizumab + Gemcitabine: Participants received bevacizumab 7.5 mg/kg IV infusion on Day 1 and gemcitabine 1200 mg/m^2 IV infusion on Days 1 and 8 of each 21-day cycle for a maximum of 6 cycles. After Cycle 6, participants continued treatment with bevacizumab 7.5 mg/kg IV infusion on Day 1 of every 21-day cycle until progressive disease, death, or intolerable toxicity.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin | Total
Number analyzed (Participants) | 44 | 42 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (3.2) | 73.8 (3.5) | 74.0 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 28 | 30 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive and Without Progressive Disease at Month 6
Description: Disease progression was assessed according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1 (v 1.1). Disease progression was defined at least a 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 millimeter (mm), progression of existing non-target lesions, or presence of new lesions.
Time Frame: Month 6
Population: Intent-to-treat (ITT) set included all participants in the RND set who received at least one dose of any study medication; participants were classified according to treatment received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 43 | 40
percentage of participants | 25.6 [12.5 to 38.6] | 30.0 [15.8 to 44.2]

2. Secondary Outcome: Percentage of Participants With Disease Progression or Death
Description: Disease progression was assessed according to RECIST criteria v1.1. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: Baseline; Day 15 of Cycles 3 and 6; Month 6 and then every 3 months until disease progression, death, or consent withdrawal (up to 53 months)
Population: ITT set
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 43 | 40
percentage of participants | 86.0 | 90.0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the interval between the date of randomization and the first documentation of progressive disease or death from any cause. Disease progression was assessed according to RECIST criteria v 1.1. Disease progression was defined at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. PFS was estimated using Kaplan Meier method.
Time Frame: as for outcome 2
Population: ITT set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 43 | 40
months | 4.33 [2.20 to 5.97] | 6.82 [4.49 to 8.52]

4. Secondary Outcome: Percentage of Participants Alive at 12 Months After Randomization
Time Frame: 1 year
Population: ITT set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 43 | 40
percentage of participants | 37.2 [22.8 to 51.7] | 47.5 [32.0 to 63.0]

5. Secondary Outcome: Percentage of Participants Who Died
Time Frame: From randomization to death or end of the study (up to 53 months)
Population: ITT set
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 43 | 40
percentage of participants | 69.8 | 72.5

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the interval between the date of randomization and death from any cause. OS was estimated using Kaplan Meier method.
Time Frame: From randomization to death or end of the study (up to 53 months)
Population: ITT set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 43 | 40
months | 5.66 [3.38 to 13.0] | 12.0 [9.93 to 19.6]

7. Secondary Outcome: Percentage of Participants by Best Overall Response
Description: Best overall response was defined as the best response recorded from the start of the treatment until disease progression/recurrence, assessed according to RECIST criteria v 1.1. Complete Response (CR): disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to less than (<) 10 millimeter (mm) in short axis; Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesion, and no new lesions; Progressive Disease (PD): at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions; Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Baseline; Day 15 of Cycles 3 and 6; Month 6 and then every 3 months until disease progression, death or consent withdrawal (up to 53 months)
Population: ITT set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 43 | 40
percentage of participants
  CR | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  PR | 14.0 [3.6 to 24.3] | 35.0 [20.2 to 49.8]
  SD | 39.5 [24.9 to 54.1] | 37.5 [22.5 to 52.5]
  PD | 16.3 [5.2 to 27.3] | 12.5 [2.2 to 22.7]
  Not Assessable | 30.2 [16.5 to 44.0] | 15.0 [3.9 to 26.1]

8. Secondary Outcome: Percentage of Participants With an Objective Response
Description: Objective response was defined as having a CR or PR according to a RECIST criteria v 1.1. CR was defined as disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions.
Time Frame: Cycle 3 Day 15, Cycle 6 Day 15 and at Month 6
Population: ITT set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 43 | 40
percentage of participants
  Cycle 3 | 11.6 [2.05 to 21.2] | 27.5 [13.7 to 41.3]
  Cycle 6 | 9.3 [0.62 to 18.0] | 15.0 [3.93 to 26.1]
  Month 6 | 4.7 [0.00 to 10.9] | 10.0 [0.70 to 19.3]

9. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease control was defined as having CR/PR/SD as per RECIST criteria v 1.1. CR was defined as disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: Cycle 3 Day 15, Cycle 6 Day 15 and at Month 6
Population: ITT set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 43 | 40
percentage of participants
  Cycle 3 | 53.5 [38.6 to 68.4] | 67.5 [53.0 to 82.0]
  Cycle 6 | 27.9 [14.5 to 41.3] | 37.5 [22.5 to 52.5]
  Month 6 | 25.6 [12.5 to 38.6] | 30.0 [15.8 to 44.2]

10. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined for participants who had achieved an objective response (CR/PR) (whichever status was recorded first) as the time period from first documentation of a response to the date of first occurrence of investigator documented disease progression or death. CR was defined as disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. Disease progression was defined as increase by at least 20% in the sum of the longest diameters of each target lesion, taking as a reference the smallest sum of the longest diameters or appearance of one or more new lesions. DoR was estimated using Kaplan Meier method.
Time Frame: as for outcome 7
Population: ITT set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 43 | 40
months | 5.23 [3.93 to NA] — It was not possible to estimate the statistic using Kaplan-Meier because upper bound of 95% confidence interval was not reached. | 5.97 [2.20 to 9.08]

ADVERSE EVENTS:
Time Frame: From baseline to 28 days after last dose of any study drug (up to 54 months)
Description: Safety set included all participants in the RND set who received at least one dose of any study medication. Participants were classified according to treatment received.
Arm/Group | Bevacizumab + Gemcitabine | Bevacizumab + Gemcitabine + Cisplatin
Serious Adverse Events (participants affected / at risk) | 17/43 | 10/40
Other Adverse Events (participants affected / at risk) | 38/43 | 37/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Gemcitabine (N=43) | Bevacizumab + Gemcitabine + Cisplatin (N=40)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0
Embolism (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Gemcitabine (N=43) | Bevacizumab + Gemcitabine + Cisplatin (N=40)
Anaemia (Blood and lymphatic system disorders) | 5 | 12
Leukopenia (Blood and lymphatic system disorders) | 0 | 11
Neutropenia (Blood and lymphatic system disorders) | 12 | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 16
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 8 | 17
Vomiting (Gastrointestinal disorders) | 5 | 6
Asthenia (General disorders) | 9 | 10
Chest pain (General disorders) | 4 | 2
Fatigue (General disorders) | 8 | 15
Mucosal inflammation (General disorders) | 0 | 5
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 8 | 8
Tooth abscess (Infections and infestations) | 0 | 2
Blood creatinine increased (Investigations) | 0 | 4
Platelet count decreased (Investigations) | 4 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness (Nervous system disorders) | 3 | 8
Paraesthesia (Nervous system disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Embolism (Vascular disorders) | 0 | 5
Hypertension (Vascular disorders) | 11 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.